CLINICAL TRIAL: NCT00808626
Title: Phase II Investigation of 99mTc-rBitistatin for Imaging Venous Thrombosis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding to complete trial. A lead member of research team retired.
Sponsor: Temple University (Other)
Responsible Party: Alan H. Maurer, MD / Director of Nuclear Medicine, Temple University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11556
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — bitistatin

ARMS (1):
- 99mTc-rBitistatin (Experimental)
  Interventions: Drug: 99mTc-rBitistatin

INTERVENTIONS:
Drug: 99mTc-rBitistatin — Intravenous administration of a single dose (10 mCi, 0.1 ug/kg body weight) of 99mTc-rBitistatin, followed by collection of scintigraphic (planar and SPECT) images at 1 hour and 2-4 hours.
  Other Names: Bitistatin; HN-Bitistatin; 99mTc-Bitis; Bitis

SUMMARY:
99mTc-rBitistatin is a radiolabeled polypeptide which is designed to stick to blood clots so that the blood clots can be detected by imaging. The purpose of this trial is to evaluate in patients the safety of 99mTc-rBitistatin and its ability to locate blood clots in the arms and legs.

ELIGIBILITY:
Inclusion Criteria:

* peripheral acute venous thrombosis diagnosed by vascular ultrasound
* is able to give informed consent
* is likely to complete the study

Exclusion Criteria:

* is pregnant
* is lactating
* has a history of prior severe allergic reactions (anaphylactic response)
* prior use of GP IIb/IIIa antagonist (e.g., abciximab, eptifibatide)
* has a platelet count <100,000 or history of thrombocytopenia
* has a history of stroke
* has a history of recent bleeding documented by decreasing hemoglobin (>1 gm) in last 7 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Establish the proof of concept that 99mTc-rBitistatin enables imaging of peripheral venous thrombi | 1-4 hours after administration

SECONDARY OUTCOMES:
Continue to evaluate the safety of 99mTc-rBitistatin administered intravenously | 0-4 hr, 6 hr, 3-4 weeks, 3-4 months after administration

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Maurer, MD, Study Director — Temple University Hospital
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States